CLINICAL TRIAL: NCT01899950
Title: Longitudinal Study of Cognition With Niemann-Pick Disease, Type C
Acronym: NPC
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Marc C. Patterson, M.D., Principal Investigator, Mayo Clinic
Other Study IDs: 11-003868; U54NS065768 (NIH); LDN6715
Record Dates: First submitted 2013-07-04; First posted 2013-07-16 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Niemann-Pick Disease, Type C
Keywords: Niemann-Pick disease type C; Lysosomal disease
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Niemann-Pick Disease, Type C (NPC) is a rare neurodegenerative disorder with a wide clinical spectrum and variable age of onset. Classically, children with NPC demonstrate neurological dysfunction with cerebellar ataxia (an inability to coordinate balance, gait, extremity and eye movements), dysarthria (difficulty speaking), seizures, vertical gaze palsy (ability to move eyes in the same direction) motor impairment, dysphagia (trouble swallowing), psychotic episodes, and progressive dementia. There is no curative treatment for NPC and it is a lethal disorder. The purpose of this protocol is to obtain both baseline and rate of progression data on a clinical and biochemical markers that may later be used as outcome measures in a clinical trial. Specifically, this study will examine and characterize the longitudinal progression of neurocognitive symptoms of NPC with the goal of identifying early markers of disease progression that may be utilized in later trials to evaluate treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

All individuals between the ages of 2 years and 99 with an established diagnosis of Niemann-Pick Disease, Type C (biochemical or molecular) will be considered for this study. Patients with both Niemann-Pick Disease, Type C1 (NPC1) and Niemann-Pick Disease, Type C2 (NPC2) mutations are eligible to participate.

Exclusion Criteria:

Participants with at least one of the following will not be eligible for this study:

1. Individuals that cannot travel because of their medical condition or are too ill to be cared for at home,
2. Individuals with stage 4 disease (non-ambulant with vegetative disturbances)
3. Individuals will be excluded if English is not their primary language

Ages: 2 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Longitudinal observational study of cognition in patients with NPC. Subjects will be recruited from participants in an observational study currently in progress at NIH, and from subjects receiving clinical care at Mayo Clinic. Participants will be administered age-and functionally-appropriate neuropsychological test instruments annually to track cognitive changes over time, and to link these data to the subjects' scores on the NIH disability scale.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2011-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Composite score of neurocognitive measures | Baseline and at yearly intervals for five years
  The composite score of neurocognitive measures will be calculated as follows: raw scores of neurocognitive tests will be transformed to Z-scores on normative data to allow comparison across measures administered at different ages. A score will be generated for each of the following domains: Intellectual Ability,Visual-Spatial Skills, Rote Verbal Memory, Narrative Verbal Memory, Visual-Spatial Construction, Nonverbal Working Memory, Language, Fine Motor, Attention, Executive Functioning, and Adaptive Behavior. Behavioral and emotional difficulties will be rated in terms of presence or absence of symptoms above a clinical cutoff score.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Patterson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States